CLINICAL TRIAL: NCT06186544
Title: Prospective Longitudinal Study To Validate Accuracy Of The Global Anatomical Staging System (GLASS) Score In Predicting Major Acute Limb Events In Patients With Chronic Limb Threatening Ischemia Undergoing Endovascular Intervention
Brief Title: Validating GLASS Score in Predicting Acute Limb Events in CLTI Patients
Acronym: PROMOTEGLASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: The European Vascular Research Collaborative (EVRC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8682; 323934 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2023-12-07; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Chronic Limb-Threatening Ischemia
Keywords: CLTI; Chronic Limb Threatening Ischemia; Revascularization; MALE; MLLA; Limb based patency; Global Anatomical Staging system (GLASS); Angioplasty; Lower limb bypass
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ischemia is a severe medical condition that occurs when the blood and oxygen supply to a specific part of the body is significantly reduced or completely absent, it can affect any body part, often the legs. It is typically caused by the narrowing or blockage of an artery and can result in severe pain, tissue gangrene, and the potential loss of a limb (Amputation). This condition requires medical intervention and will not improve on its own.

To diagnose leg ischemia, the doctor will conduct a thorough vascular clinical examination. Depending on the findings, further imaging tests such as duplex ultrasound, magnetic resonance arteriography (MRA), or computed tomography (CT) may be conducted. In some cases, an arteriogram may be necessary which is an x-ray of the arteries while the dye is injected into the blood vessels.

Following the diagnosis, the best management course is recommended by a multidisciplinary team (MDT), considering each patient's disease pattern and overall health. Treatment options include performing a key-hole procedure, called an endovascular procedure (EVT) within the artery, where the vascular surgeon will be using a balloon to widen the artery, and/or a wire-reinforced stent which remains inside the artery serving as a scaffolding to keep it open.

The primary aim of the PROMOTE GLASS study is to investigate if the Global Anatomical Staging System (GLASS) score, which is a summation of points given according to the disease pattern as seen on assessment images (Duplex Ultrasound, MRA, and CT scans) can accurately tell if the treatment using catheters and stents inside blood vessels will work well for people with ischemia in their legs. The researchers also want to see if the GLASS score can predict how well patients with ischemia will heal and if they will need further treatments in the long term after having treatment with catheters and stents inside their blood vessels.

A prospective, observational study will be delivered by Cardiff and Vale University Health Board (CAVUHB). The vascular team will prospectively collect data over a 12-month period. This will be in patients undergoing elective and/or emergency primary EVT procedure, with follow-up 4-6 weeks after the procedure and at 12 months.

DETAILED DESCRIPTION:
The Global Vascular Guideline (GVG) is an expert consensus, representing every major vascular society, aiming to promote a standardized evidence-based approach to assessing and treating patients with Chronic Limb Threatening Ischemia (CLTI). In terms of revascularization, the GVG recommendations revolve around three independent variables: patient risk, limb severity, and anatomic complexity (PLAN). Each section is fundamental to providing successful treatment to the patient, much controversy remains on which patterns of anatomical disease should be treated with endovascular or open surgery. To that end, the GLobal Anatomic Staging System (GLASS) was developed and adopted by the GVG committee as an angiographic scoring system to quantify the extent of infra-inguinal disease and predict the likely success of treatment with endovascular techniques (EVT).

GLASS is intended to predict the immediate technical success (ITS) and the 1-year limb base patency (LBP) after the EVT of the target artery pathway (TAP) and therefore aid in decision making. Currently there is no other risk prediction score or risk prediction model that estimates the probability of having ITS, LBP, major adverse limb events (MALE), major lower limb amputation (MLLA) and overall survival (OS) in patients presenting with CLTI who undergo EVT.

The purpose of this longitudinal prospective study is to examine the validity and reliability of the GLASS score in predicting ITS, LBP, MALE, MLLA, and OS in patients with CLTI, eventually helping to identify those patients who are likely to benefit from EVT. This could help clinicians make more informed decisions about treatment options, potentially reducing the need for more invasive procedures and improving patient outcomes. Additionally, the GLASS score could be used as a tool for patient selection in future clinical trials evaluating endovascular interventions for CLTI.

This study will follow a prospective observational study design. The study will initially be conducted within the Southeast Wales Vascular Network at Cardiff and Vale University Health Board. However, the study protocol allows for the inclusion of other hospitals or vascular units to participate in a collaborative model or as primary investigator sites, subject to obtaining necessary ethics approval and sponsorship agreement. The decision to involve additional sites will be made following a thorough evaluation by the research and development (R&D) committee. This approach will ensure compliance with ethical guidelines and regulatory requirements while also fostering potential collaboration and broadening the study's reach and generalizability.

Patients will be identified through routine clinic referrals and emergency presentations with CLTI; only patients who are referred for EVT will be recruited. Recruited patients will consent to access to their medical files and radiological data (duplex scans and angiography images) and a clinical follow-up up to one year. Standard care pathways are followed beyond this point. Outcome data will be collected from patients' medical files and interventional radiology reports immediately after the EVT and from vascular surgery clinic follow-up notes over a 12 months period. Symptom scores, admissions records, clinical and imaging data will be analysed at the end of follow-up to validate risk prediction. This will be supported by the European Vascular Research Collaborative (EVRC).

This study will be supervised by the Chief Investigator, Mr. Lewis Meecham (Consultant Vascular and Endovascular Surgeon) and sponsored by Cardiff and Vale University Health Board. An internal management group consisting of clinicians, researchers and managerial staff will be established to oversee and monitor the progress of the study. The management group will meet on a monthly basis to raise, discuss, and resolve any issues arising during the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral vascular disease (PVD) under investigation for CLTI
2. Age 18 years or older
3. Able to consent to inclusion.

Exclusion Criteria:

1. Patient with traumatic or iatrogenic lesions leading to CLTI.
2. Acute Limb Ischemia (symptoms for <2 weeks)
3. Patients who have undergone open/endovascular revascularization of the same limb within the last 12 months
4. Patients who present with inflow disease (Common iliac artery (CIA), External Iliac Artery (EIA), and Common Femoral artery (CFA) disease) not intended for treatment during the same admission or prior to recruitment.
5. Palliative revascularization (for pain in end of life)
6. Patient with expected problems of maintaining a 1-year follow-up (e.g., no fixed address)
7. Patients with previously implanted devices (stents) within the affected segment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will consist of adult vascular patients diagnosed with chronic limb threatening ischemia (CLTI) who are scheduled to undergo endovascular intervention according to the standard care pathway. These participants will be selected from vascular surgery MDT and will represent a diverse range of demographics and clinical characteristics. Participants will be included based on specific eligibility criteria, such as age, severity of CLTI, previous interventions in the limb of interest and willingness to participate in the study. Throughout the study, participants will be followed longitudinally, with their GLASS scores recorded at presentation and major acute limb events monitored over 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Immediate Technical Success i.e. achievement of straight in-line flow to the foot as judged from the completion angiography | Day 0
  Immediate technical success (ITS): The successful completion of endovascular therapy procedures without any major complications. Specifically, it is the successful achievement of the intended treatment goals, such as revascularization, stent deployment, or atherectomy. A procedure is considered to have achieved ITS when the desired therapeutic objectives are accomplished and the patient's vascular anatomy is adequately restored, without the need for additional intervention or conversion to open surgery.
Rate of The immediate technical failure (ITF) | Day 0
  Immediate technical failure (ITF): ITF is defined as the inability to successfully perform the desired endovascular intervention due to technical limitations. It encompasses scenarios such as inadequate vessel access, equipment malfunction, or procedural complications that prevent the completion of the intended procedure.
Rate of LBP (as judged by the main surgeon based on symptoms and imaging up to 12 months) | Day 1 and up to 12 months
  Limb based patency (LBP): limb-based patency (LBP) is defined as continued patency throughout the length of a defined target artery pathway (TAP) from the groin to the ankle.
  The TAP consists of the femoropopliteal (FP) segment, and a primary infrapopliteal (IP) runoff artery selected by the treating physician to achieve in-line flow to the foot or wound. LBP combines freedom from reintervention, occlusion, and severe stenosis of the TAP, along with freedom from hemodynamic failure (a significant decrease in ankle or toe pressures) in the presence of recurrent or unresolved CLTI symptoms.

SECONDARY OUTCOMES:
Rate of MALE (as judged by the main surgeon based on symptoms and imaging up to 12 months) | Day 1 and up to 12 months
  Major adverse limb events (MALE): MALE is defined as limb-related events including major amputations, acute limb ischemia requiring urgent revascularization, or repeat interventions due to disease progression or complications.
Rate of MLLA (as judged by the main surgeon based on symptoms and imaging up to 12 months) | Day 1 and up to 12 months
  Major Lower Limb Amputation (MLLA): MLLA is defined as above ankle amputations of the leg i.e. either above knee amputation (Transfemoral amputation), below knee amputation (Transtibial amputation), or through knee amputation.
Overall survival (in months) | Day 1 and up to 12 months
  Overall survival (OS): OS is defined as freedom from death up to 12 months from the treatment date due to any cause.
Timings of any adverse clinical event (MALE, MLLA, Mortality) | Day 1 and up to 12 months
  If presented before the scheduled follow up

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Meecham, FRCS, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- Southeast Wales Vascular Network-Cardiff and Vale University Health Board, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study will take place in Cardiff and Vale UHB. All investigators and researchers must comply with the requirements of the General Data Protection Regulation (GDPR) Europe (EU) (2016/679) with regards to the collection, storage, processing, and disclosure of personal information.
  Data collected during the course of the study will be kept strictly confidential and accessed only by members of the study team. Data will be entered directly into the study database via a secure data capture and management software (CASTOR) that is GDPR compliant, access will be granted for the responsible surgeons only. Each case will be given a pseudo-anonymized number to avoid sharing of patient identifiable information.
  Study data will be archived in accordance with the Cardiff & Vale UHB Archiving of Clinical Trial and Research Study Data Standard Operating Procedure. No personal identifiable data relating to patients will be retained beyond the end of the study.

REFERENCES:
- [Derived] Darwish M, D'Oria M, Croo A, Melo RG, Meecham L; European Vascular Research Collaborative (EVRC). Prospective Multi-Center Longitudinal Study to Validate Accuracy of the Global Anatomic Staging System (GLASS) Score in Predicting Major Acute Limb Events in Patients With Chronic Limb Threatening Ischemia Undergoing Endovascular Intervention: The PROMOTE-GLASS Study Protocol. Vasc Endovascular Surg. 2025 Jan;59(1):29-38. doi: 10.1177/15385744241276690. Epub 2024 Sep 3. PMID 39226237